CLINICAL TRIAL: NCT00561821
Title: A Double-Blind, Randomized, Parallel Group, Placebo- Controlled Sleep Laboratory Efficacy and Safety Study With Org 50081 in Elderly Subjects With Chronic Primary Insomnia
Brief Title: Efficacy and Safety Study of Org 50081 (Esmirtazapine) in Elderly Participants (P05709)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05709; 21108 (Other: Organon); MK-8265-006 (Other: Merck Study Number)
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Insomnia; Sleep Initiation and Maintenance Disorders; Mental Disorders; Dyssomnias; Sleep Disorders
Keywords: elderly; randomized; placebo controlled
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Mental Disorders; Dyssomnias; Sleep Wake Disorders | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Esmirtazapine 0.5 mg (Experimental): one placebo tablet daily for 14 days, followed by one 0.5 mg tablet Esmirtazapine daily for 16 days, and then one placebo tablet daily for 7 days
  Interventions: Drug: Esmirtazapine; Drug: Placebo
- Esmirtazapine 1.5 mg (Experimental): one placebo tablet daily for 14 days, followed by one 1.5 mg tablet Esmirtazapine daily for 16 days, and then one placebo tablet daily for 7 days
  Interventions: Drug: Esmirtazapine; Drug: Placebo
- Esmirtazapine 3.0 mg (Experimental): one placebo tablet daily for 14 days, followed by one 3.0 mg tablet Esmirtazapine daily for 16 days, and then one placebo tablet daily for 7 days
  Interventions: Drug: Esmirtazapine; Drug: Placebo
- Placebo (Placebo Comparator): one placebo tablet daily for 14 days, followed by one placebo tablet daily for 16 days, and then one placebo tablet daily for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esmirtazapine — one tablet daily
  Arms: Esmirtazapine 0.5 mg; Esmirtazapine 1.5 mg; Esmirtazapine 3.0 mg
Drug: Placebo — one tablet daily

SUMMARY:
This study was conducted to investigate the efficacy of treatment with Org 50081 (Esmirtazapine)

compared to placebo in elderly participants with chronic primary

insomnia. Primary efficacy variable is Wake time After Sleep

Onset (WASO), averaged over all in-treatment time points

and measured by polysomnography (PSG).

DETAILED DESCRIPTION:
Insomnia is a common complaint or disorder throughout the

world. About one third of the population in the industrial

countries reports difficulty initiating or maintaining sleep,

resulting in a non-refreshing or non-restorative sleep. The

majority of the insomniacs suffer chronically from their

complaints.

The maleic acid salt of Org 4420, code name Org 50081, known as Esmirtazapine, was

selected for development in the treatment of insomnia. The

first clinical trial with Esmirtazapine was a proof-of-concept trial

with a four-way cross-over design. All 3 Esmirtazapine dose

groups showed a statistically significant positive effect on

TST (objective and subjective) and WASO, as compared to

placebo.

The current study is designed to assess the efficacy and safety

of Esmirtazapine in a double-blind, placebo-controlled, parallel,

randomized trial in elderly participants suffering from chronic

primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* are at least 65 years of age at screening;
* sign written informed consent after the scope and

nature of the investigation have been explained to

them, before screening evaluations;

* are able to speak, read and understand the language of

the investigator, study staff (including raters) and the

informed consent form, and possess the ability to

respond to questions, follow instructions and complete

questionnaires;

* have demonstrated capability to independently

complete the LogPad questionnaires and have

completed the questionnaires at least 6 out of 7 days of

the week preceding randomization;

* have a regular sleep pattern, meaning bedtime regularly

occurs between 2100 hours and 2400 hours, with no more variation

from these boundaries than 2 times/ week, with 5-8.5

hours in bed;

* have a documented diagnosis of chronic primary

insomnia, defined as fulfillment of the Diagnostic and Statistical Manual of Mental Disorders IV - Text Revision (DSM-IV-TR) criteria

for primary insomnia (DSM-IV-TR 307.42) with a duration

of >= 1 month; fulfill the following PSG criteria on the

two screening/baseline PSG nights:

* average Total Sleep Time (TST) < 6.5 h (and each night greater than or

equal to 3 h and < 7 h),

* average WASO greater than or equal to 45 minutes

(and each night greater than or equal to 30 min),

* average Latency to Persistent Sleep (LPS) 15 min (and each night greater than or

equal to 10 min).

Exclusion Criteria:

* have other sleep disorders (DSM-IV-TR), such as sleep

related breathing disorders Apnea-Hypopnea Index (AHI) greater than or equal

to 15), Periodic Leg Movements with Arousals Index (PLMAI)

greater than or equal to 10), restless leg syndrome,

narcolepsy, circadian sleep wake rhythm disorders,

Rapid Eye Movement (REM) behavioral disorder or any parasomnia;

* have any significant medical or DSM-IV-TR

psychiatric illness causing the sleep disturbances;

* currently meet diagnostic criteria for DSM-IV-TR

depression Major Depressive Disorder (MDD) or have been diagnosed and treated

for MDD within the last 2 years;

* have a history of bipolar disorder, a history of suicide attempt or a family history of suicide. A family history of suicide is defined as any history of suicide in the first and second degree family (parents, siblings, grandparents, or offspring), or a pattern of completed suicides (more than one) in the third degree family (aunts, uncles, nieces and nephews);
* have a history or signs of dementia or other serious

cognitive impairment, as defined by a score of less than

26 on the Mini-Mental State Examination;

* have a significant, unstable medical illness e.g. acute or

chronic pain, hepatic, renal, metabolic or cardiac

disease;

* had serious head injury or stroke within the past year,

or a history of (non-febrile) seizures;

* have clinically relevant electrocardiogram (ECG) abnormalities at

screening, as judged by the investigator;

* have clinically relevant abnormal hematology or

biochemistry values at screening, as judged by the

investigator;

* have DSM-IV-TR substance abuse or DSM-IV-TR

addiction within the last year;

* drink more than 2 alcoholic drinks in a day. One drink is approximately equal to: 12 oz or 360 ml of beer (regular or light), or 4 oz or 120 ml of red or white wine, or 2 oz or 60 ml of desert wine (e.g. port, sherry), or 12 oz or 360 ml of wine cooler (regular or light), or 1 oz or 30 ml or spirits (80 to 100 proof, e.g. whiskey, vodka);
* are routinely sleeping during daytime (napping) for more than 20 minutes per day, 3 days or more per week;
* are night workers or rotating shift workers currently, or in the past 6 months
* use of psychotropic drugs affecting sleep within two weeks prior to randomization (fluoxetine: five weeks);
* use of concomitant medication affecting sleep (e.g. anxiolytics, sedatives, antidepressants, antipsychotics, centrally active sedating antihistamines, central nervous system (CNS)

stimulants, alpha-2-antagonists, respiratory stimulants and decongestants);

* smoke > 15 cigarettes per day and/or can not abstain from smoking during the night;
* drink excessive amounts of caffeinated beverages/day (more than 500 mg caffeine per day);
* have a body mass index (BMI) >= 36;
* have a positive urine drug screen at screening or at baseline;
* have a known hypersensitivity to mirtazapine or to any of the excipients;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 538 (Actual)
Dates: Start 2007-11-20 (Actual); Primary Completion 2009-12-21 (Actual); Study Completion 2009-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Esmirtazapine 0.5 mg: One placebo tablet daily for 14 days, followed by a double-blind treatment period of one 0.5 mg tablet Esmirtazapine daily for 16 days, and then one placebo tablet daily for 7 days
- Esmirtazapine 1.5 mg: One placebo tablet daily for 14 days, followed by a double-blind treatment period of one 1.5 mg tablet Esmirtazapine daily for 16 days, and then one placebo tablet daily for 7 days
- Esmirtazapine 3.0 mg: One placebo tablet daily for 14 days, followed by a double-blind treatment period of one 3.0 mg tablet Esmirtazapine daily for 16 days, and then one placebo tablet daily for 7 days
- Placebo: One placebo tablet daily for 14 days, followed by a double-blind treatment period of one placebo tablet daily for 16 days, and then one placebo tablet daily for 7 days
Period: Overall Study
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Started | 132 | 136 | 134 | 136
Treated | 132 | 136 | 133 | 136
Completed | 127 | 130 | 132 | 133
Not Completed | 5 | 6 | 2 | 3
Not completed — Not treated | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2
Not completed — Reasons not related to trial | 2 | 1 | 0 | 0
Not completed — Other (reason not specified) | 1 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All Subjects Treated (AST) population consisted of participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo | Total
Number analyzed (Participants) | 132 | 136 | 133 | 136 | 537
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.1 (4.4) | 70.0 (4.4) | 71.1 (4.6) | 70.3 (4.3) | 70.4 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 82 | 88 | 82 | 336
  Male | 48 | 54 | 45 | 54 | 201

OUTCOME MEASURES:

1. Primary Outcome: Average Wake Time After Sleep Onset Measured by Polysomnography
Description: Wake time after sleep onset (WASO) is the total time awake between sleep onset and "lights on"; i.e. from the onset of persistent sleep until the end of the 8-hour polysomnography (PSG) recording. PSG assesses the quality of sleep by monitoring brain waves, breathing, heart function, muscle activity and eye movement. PSG measurements of WASO (observed data only) taken during the 16-day double-blind treatment period, over days 1 and 2 and days 15 and 16, were averaged.
Time Frame: Up to Day 16
Population: The intent to treat (ITT) population consisted of all randomized participants who received at least one dose of double-blind study medication and had at least one post-randomization efficacy assessment. Data from 11 participants located at one treatment site were not analyzed due to their lack of credibility.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 133
Minutes | 80.3 (36.5) | 79.6 (30.7) | 74.8 (28.0) | 109.8 (42.1)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Pairwise comparisons on rank transformed data with effects for treatment and center, and baseline of variable as a covariate
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Average Latency to Persistent Sleep Measured by Polysomnography
Description: Latency to Persistent Sleep (LPS) is the time from lights out to the first 20 consecutive epochs scored as sleep by PSG. PSG assesses the quality of sleep by monitoring brain waves, breathing, heart function, muscle activity and eye movement. PSG measurements of LPS (observed data only) taken during the 16-day double-blind treatment period, over days 1 and 2 and days 15 and 16, were averaged.
Time Frame: Up to Day 16
Population: The ITT population consisted of all randomized participants who received at least one dose of double-blind study medication and had at least one post-randomization efficacy assessment. Data from 11 participants located at one treatment site were not analyzed due to their lack of credibility.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 133
Minutes | 32.3 (24.8) | 30.7 (23.0) | 29.3 (22.8) | 37.1 (25.7)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.0146, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p = 0.0234, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.0102, ANCOVA — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Average Total Sleep Time Measured by Polysomnography
Description: Total sleep time (TST) is the sleep time recorded by PSG. PSG assesses the quality of sleep by monitoring brain waves, breathing, heart function, muscle activity and eye movement. PSG measurements of TST (observed data only) taken during the 16-day double-blind treatment period, over days 1 and 2 and days 15 and 16, were averaged.
Time Frame: Up to Day 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 133
Minutes | 374.1 (39.9) | 376.2 (34.9) | 383.4 (35.7) | 338.7 (45.8)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Average Number of Awakenings Measured by Polysomnography
Description: Number of awakenings (NAW) was measured by PSG. PSG assesses the quality of sleep by monitoring brain waves, breathing, heart function, muscle activity and eye movement. PSG measurements of NAW (observed data only) taken during the 16-day double-blind treatment period, over days 1 and 2 and days 15 and 16, were averaged.
Time Frame: Up to Day 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of awakenings
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 133
Number of awakenings | 13.5 (5.4) | 13.4 (4.7) | 13.5 (4.7) | 12.1 (4.8)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p = 0.0213, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.0135, ANCOVA — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Average Wake Time After Sleep Onset in the First Quarter of the Night Measured by Polysomnography
Description: Wake time after sleep onset (WASO) is the total time awake between sleep onset and "lights on"; i.e. from the onset of persistent sleep until the end of the 8-hour PSG recording. WASO was recorded in the first quarter of the night, for at most 2 hours, by PSG. PSG assesses the quality of sleep by monitoring brain waves, breathing, heart function, muscle activity and eye movement. PSG measurements of WASO (observed data only) taken during the 16-day double-blind treatment period, over days 1 and 2 and days 15 and 16, were averaged.
Time Frame: Up to Day 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 133
Minutes | 34.5 (17.4) | 33.7 (16.2) | 31.2 (15.6) | 40.6 (20.0)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Average Wake Time After Sleep Onset in the Second Quarter of the Night Measured by Polysomnography
Description: Wake time after sleep onset (WASO) is the total time awake between sleep onset and "lights on"; i.e. from the onset of persistent sleep until the end of the 8-hour PSG recording. WASO was recorded in the second quarter of the night, for at most 2 hours, by PSG. PSG assesses the quality of sleep by monitoring brain waves, breathing, heart function, muscle activity and eye movement. PSG measurements of WASO (observed data only) taken during the 16-day double-blind treatment period, over days 1 and 2 and days 15 and 16, were averaged.
Time Frame: Up to Day 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 133
Minutes | 20.1 (11.7) | 19.2 (11.4) | 18.9 (10.4) | 25.9 (13.7)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Average Wake Time After Sleep Onset in the Third Quarter of the Night Measured by Polysomnography
Description: Wake time after sleep onset (WASO) is the total time awake between sleep onset and "lights on"; i.e. from the onset of persistent sleep until the end of the 8-hour PSG recording. WASO was recorded in the third quarter of the night, for at most 2 hours, by PSG. PSG assesses the quality of sleep by monitoring brain waves, breathing, heart function, muscle activity and eye movement. PSG measurements of WASO (observed data only) taken during the 16-day double-blind treatment period, over days 1 and 2 and days 15 and 16, were averaged.
Time Frame: Up to Day 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 133
Minutes | 20.5 (12.0) | 21.3 (11.6) | 19.1 (10.4) | 31.9 (18.5)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Average Wake Time After Sleep Onset in the Fourth Quarter of the Night Measured by Polysomnography
Description: Wake time after sleep onset (WASO) is the total time awake between sleep onset and "lights on"; i.e. from the onset of persistent sleep until the end of the 8-hour PSG recording. WASO was recorded in the fourth quarter of the night, for at most 2 hours, by PSG. PSG assesses the quality of sleep by monitoring brain waves, breathing, heart function, muscle activity and eye movement. PSG measurements of WASO (observed data only) taken during the 16-day double-blind treatment period, over days 1 and 2 and days 15 and 16, were averaged.
Time Frame: Up to Day 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 133
Minutes | 30.9 (17.6) | 29.7 (13.5) | 27.4 (14.9) | 42.4 (23.2)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Average Number of Stage Shifts to Stage 1 or Wake Measured by Polysomnography
Description: Number of stage shifts to stage 1 of sleep or to awaken was measured by PSG. A stage shift is the transition measured by PSG between various sleep stages. PSG assesses the quality of sleep by monitoring brain waves, breathing, heart function, muscle activity and eye movement. PSG measurements of the number of stage shifts (observed data only) taken during the 16-day double-blind treatment period, over days 1 and 2 and days 15 and 16, were averaged.
Time Frame: Up to Day 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of stage shifts
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 133
Number of stage shifts | 51.8 (16.0) | 50.6 (15.3) | 51.3 (16.1) | 44.0 (15.7)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Average Subjective Total Sleep Time Based on Sleep Diary
Description: Total Sleep Time (TST) is a subjective time (observed data only) recorded daily by the participant in an electronic diary, that was averaged over the entire 16-day, double-blind treatment period.
Time Frame: Up to Day 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 132
Minutes | 364.4 (61.4) | 357.3 (73.2) | 368.8 (63.9) | 339.9 (52.7)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

11. Secondary Outcome: Average Subjective Sleep Latency Based on Sleep Diary
Description: Sleep latency (SL) is the time taken to fall asleep (observed data only) recorded daily by the participant in an electronic diary, that was averaged over the entire 16-day, double-blind treatment period.
Time Frame: Up to Day 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 132
Minutes | 51.6 (48.9) | 53.1 (39.9) | 50.5 (43.0) | 46.5 (26.3)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.6317, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p = 0.6355, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.7865, ANCOVA — [p-value comment as in outcome 1, analysis 1]

12. Secondary Outcome: Average Subjective Number of Awakenings Based on Sleep Diary
Description: Number of awakenings between sleep onset and final awakening (NAW) is a subjective number (observed data only) recorded daily by the participant in an electronic diary, that was averaged over the entire 16-day, double-blind treatment period.
Time Frame: Up to Day 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of Awakenings
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 132
Number of Awakenings | 1.9 (1.2) | 2.2 (1.8) | 2.1 (1.3) | 1.9 (1.0)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.4033, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p = 0.4153, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.6271, ANCOVA — [p-value comment as in outcome 1, analysis 1]

13. Secondary Outcome: Average Subjective Wake Time After Sleep Onset Based on Sleep Diary
Description: Wake Time after Sleep Onset (WASO) is after falling asleep initially, the subjective time that the participant was awake during the night. Daily recordings by the participant in an electronic diary (observed data only), were averaged over the entire 16-day, double-blind treatment period.
Time Frame: Up to Day 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 132
Minutes | 58.4 (38.9) | 70.3 (53.1) | 62.2 (45.4) | 81.7 (50.0)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]

14. Secondary Outcome: Average Subjective Quality of Sleep Based on Sleep Diary
Description: Quality of Sleep (QS) is a subjective number on a Visual Analog Scale ranging from 0 to 100, where very poor is rated at 0, up to excellent, rated at 100. Daily recordings by the participant in an electronic diary (observed data only) were averaged over the entire 16-day, double-blind treatment period.
Time Frame: Up to Day 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 132
Units on a Scale | 57.8 (16.1) | 56.7 (17.0) | 58.0 (17.4) | 54.8 (18.1)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.0243, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p = 0.0242, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.0007, ANCOVA — [p-value comment as in outcome 1, analysis 1]

15. Secondary Outcome: Average Subjective Satisfaction of Sleep Duration Based on Sleep Diary
Description: Satisfaction of Sleep Duration (SSD) is a subjective number on a Visual Analog Scale ranging from 0 to 100, where very unsatisfied is rated at 0, up to fully satisfied, rated at 100. Daily recordings by the participant in an electronic diary (observed data only) were averaged over the entire 16-day, double-blind treatment period.
Time Frame: Up to Day 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 129 | 132 | 131 | 132
Units on a Scale | 57.8 (16.0) | 56.8 (16.4) | 58.1 (17.2) | 54.0 (17.0)
Statistical Analysis 1: Comparison: Esmirtazapine 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.0199, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Esmirtazapine 1.5 mg vs Placebo; Test type: Superiority or Other; p = 0.0316, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Esmirtazapine 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.0014, ANCOVA — [p-value comment as in outcome 1, analysis 1]

16. Secondary Outcome: Number of Participants With an Adverse Event During the 16 Day, Double-blind Treatment Period
Description: An Adverse Event (AE) is any untoward occurrence in a participant who is administered any pharmaceutical product, and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding) symptom, or disease temporarily associated with the use of an investigational medicinal product (IMP), whether or not it is related to the IMP.
Time Frame: Up to Day 16
Population: All participants who received at least one dose of study medication.
Measure: Number; unit: Number of participants
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 132 | 136 | 133 | 136
Number of participants | 48 | 54 | 56 | 40

17. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to an Adverse Event During the 16 Day, Double-blind Treatment Period
Description: An AE is any untoward occurrence in a participant who is administered any pharmaceutical product, and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding) symptom, or disease temporarily associated with the use of an IMP, whether or not it is related to the IMP.
Time Frame: Up to Day 16
Population: All participants who received at least one dose of study medication.
Measure: Number; unit: Number of participants
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Number analyzed (Participants) | 132 | 136 | 133 | 136
Number of participants | 2 | 3 | 1 | 1

ADVERSE EVENTS:
Description: Participants who received at least one dose of study medication. One of the 538 enrolled participants was not treated.
Arm/Group | Esmirtazapine 0.5 mg | Esmirtazapine 1.5 mg | Esmirtazapine 3.0 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/136 | 0/133 | 0/136
Other Adverse Events (participants affected / at risk) | 18/132 | 21/136 | 27/133 | 8/136
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmirtazapine 0.5 mg (N=132) | Esmirtazapine 1.5 mg (N=136) | Esmirtazapine 3.0 mg (N=133) | Placebo (N=136)
Fatigue (General disorders) | 7 (7) | 8 (8) | 9 (9) | 3 (3)
Dizziness (Nervous system disorders) | 9 (9) | 6 (6) | 8 (9) | 3 (3)
Somnolence (Nervous system disorders) | 6 (6) | 12 (13) | 16 (16) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less